CLINICAL TRIAL: NCT05315375
Title: Post-trauma Lumbar Vertebral Body Reconstruction Using Expandable Cages: Comprehensive Long-term Follow-up Outcomes
Brief Title: Post-trauma Lumbar Vertebral Body Reconstruction Using Expandable Cages
Status: Completed | Type: Observational
Sponsor: Centre de l'arthrose, Paris (Other)
Responsible Party: Sponsor
Other Study IDs: vlift
Record Dates: First submitted 2022-03-30; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Disc Degeneration
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Corpectomy: surgical procedure using expandable cage
  Interventions: Device: corpectomy

INTERVENTIONS:
Device: corpectomy — vertebral corpectomy using expandable cage

SUMMARY:
INTRODUCTION

The expandable cage technology is not new, but several questions remain under-studied. Among them, there are the sagittal balance, the subsidence and the adjacent disc degeneration. Moreover, assessment of the correction and kyphosis regardless of the physiological angles can possibly lead to calculation bias.

The objective of this study was to assess the extent to which the functional outcomes were correlated to the quality of the reduction, within a homogeneous series of lumbar vertebral body reconstruction with expandable cages for trauma.

MATERIAL AND METHODS Twenty-seven patients with a mean follow-up of 3.9 years were retrospectively analyzed. The Oswestry Disability Index (ODI) was the main outcome and its association with other variables was sought. The local kyphosis and the regional traumatic angle using Stagnara's physiological angles were measured. The lumbar lordosis (LL) was compared to the Pelvic Incidence (PI). The subsidence of the cage and the adjacent disc degeneration (using the UCLA grading score) were quantified. Bone quality was assessed through the Hounsfield Unit of the vertebral body.

ELIGIBILITY:
Inclusion Criteria:

* All patients suffered from a traumatic lumbar fracture requiring a posterior fusion first

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients suffered from a traumatic lumbar fracture requiring a posterior fusion first
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2010-01-02 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) | 4 years
  specific lumbar surgery score

CONTACTS AND LOCATIONS:
Overall Officials: cedric maillot, Study Director — APHP

IPD SHARING:
Plan to Share IPD: No